CLINICAL TRIAL: NCT04289948
Title: Assessing the Efficacy of Anti-staphylococcal Phages in the Management of Infected Foot Ulcers in Diabetes
Acronym: PDFI
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Funding issues meant that development of the study was halted.
Sponsor: University Hospitals of Derby and Burton NHS Foundation Trust (Other)
Collaborators: Wellcome Trust (Other); BioPhage Theraputics Limited (Unknown); Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DHRD/2018/080
Record Dates: First submitted 2018-09-03; First posted 2020-02-28 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Diabetes; Diabetic Foot; Diabetic Foot Infection
Keywords: Diabetes; Diabetic Foot Disease; Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Foot

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Work Package 1: Observational cohort pilot safety study Work Package 2: Randomised, double-blind, placebo controlled pilot study Work Package 3: Observer-blind pilot RCT
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phage (Experimental)
  Interventions: Drug: Phage
- Placebo (Placebo Comparator)
  Interventions: Drug: Phage

INTERVENTIONS:
Drug: Phage — The studies will be undertaken using a cocktail of at least 2-3 anti-staphylococcal phages produced by Intralytix Inc, Baltimore, Maryland, USA. The phages will be included in a gel designed for application directly to the wound surface and packaged in 5 ml single use tubes.

SUMMARY:
Work Package 1: Observational cohort pilot safety study Work Package 2: Randomised, double-blind, placebo controlled pilot study Work Package 3: Observer-blind pilot RCT

DETAILED DESCRIPTION:
Work Package 1

WP1 is a safety cohort pilot study targeting patients with DFU which are non-infected as determined by the IDSA criteria. 20 participants will be recruited from Diabetic Foot Clinic at the Royal Derby Hospital. Phage gel will be applied to the index ulcer after the first and second sets of measures at baseline, weeks 1, 2 and 3. Samples will be taken at baseline and weekly up to 4 weeks by surface swab and deep tissue sample for determination of bacterial colonisation using both conventional and genotypic (molecular) microbiological methods, prior to any IMP application.

Work Package 2

WP2 is a pilot double blind, placebo-controlled, randomised study targeting patients with mild or moderate infection of DFUs and comparing systemic antibiotic therapy plus phage gel against systemic antibiotics therapy plus placebo gel. A total of 50 participants from two centres (foot clinics at Royal Derby Hospital and City Campus, Nottingham University Hospitals NHS Trust) will be recruited. Phage gel or placebo will be applied to the index ulcer after the first and second sets of measures at baseline, weeks 1, 2 and 3. Samples will be taken at baseline and weekly up to 4 weeks by surface swab and deep tissue sample for determination of bacterial colonisation using both conventional and genotypic (molecular) microbiological methods

Work Package 3

WP3 is an observer-blind RCT targeting patients with mild diabetic foot infection by IDSA criteria and comparing phage gel with systemic antibiotics. A total of 50 participants from two centres (foot clinics at Royal Derby Hospital and City Campus, Nottingham University Hospitals NHS Trust) will be recruited. Those with moderately severe infections will be withheld from this work package because of the clinical and ethical issues associated with withholding antibiotics in those with a moderately severe infection.

ELIGIBILITY:
Inclusion Criteria:

1. Diabetes Mellitus according to WHO criteria
2. are aged 18 years or over
3. Additionally, patients must meet one of the following criteria to participate in the described Work Package:

   * Patients are only eligible for WP1 if they also have one or more DFUs (area 25mm2) below the malleoli without infection according to IDSA criteria that have been present for at least 4 weeks
   * Patients are only eligible for WP2 if they also have one or more DFUs (area 25mm2) below the malleoli with mild or moderate infection according to IDSA criteria that have been present for at least 4 weeks
   * Patients are only eligible for WP3 if they also have one or more DFUs (area 25mm2) below the malleoli with mild infection according to IDSA criteria that have been present for at least 4 weeks

Exclusion Criteria:

We will exclude patients who meet ANY of the following criteria:

1. with mental incapacity to give informed consent,
2. who have other major co-morbidities, which in the opinion of the investigator would mean that the patient would not be able to complete the study
3. with significant peripheral arterial disease (PAD): ABPI (ankle brachial pressure index) <0.7,
4. Who have osteomyelitis defined by agreed clinical criteria
5. who are receiving treatment with systemic glucocorticoids or other immunosuppressants,
6. who have received systemic or topical antibiotics in the preceding 14 days,
7. who are judged to require parenteral administration of antibiotics,
8. Who have been previously recruited to an earlier part of the project
9. who are women of childbearing age who are at risk of conception
10. History of antibiotic hypersensitivity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Work Package 1: To assess the safety of the use of anti-staphylococcal phages therapy on the wound bacterial microbiome of uninfected DFU's. | 7 months
  - Safety : Clinically significant change in safety bloods, vital signs, Full Blood Count (FBC), renal function, C-Reactive protein (CRP), Liver function Tests (LFT)s, Adverse events
Work Package 2 | 16 months
  To compare the effect on the microbiome of empirical systemic antibiotic therapy alone (ESAT) versus ESAT plus phage therapy in ulcers complicated by mild or moderate infection as assessed by IDSA criteria
Work Package 3 | 16 months
  To compare the use of empirical systemic antibiotic therapy versus phage therapy in ulcers complicated by mild infection on the eradication of the infection as assessed by IDSA criteria.

SECONDARY OUTCOMES:
Work Package 1: Safety of phage gel and overt toxic effect of phage gel. | 7 months
  The following outcomes will be recorded at weekly intervals for 4 weeks from baseline:
  1. Incidence of new infection
  2. Number of days of antibiotic usage
  3. Change in surface microbiome
  4. Adverse events
  5. Change in safety bloods, vital signs, FBC, renal function, CRP, LFTs
  6. Wound status (clinical infection, area, depth, extent of surface slough, pain by VAS, peri ulcer appearance)
  7. Patient well-being using a Visual Analogue Scale, 0-100mm.
  8. Vital signs (Resting pulse and blood pressure (BP))
Work Package 1: • Impact on the bacterial microbiome of anti-staphylococcal phage gel and systemically chosen antibiotics. | 7 months
  The following outcomes will be recorded at weekly intervals for 4 weeks from baseline:
  1. Incidence of new infection
  2. Number of days of antibiotic usage
  3. Change in surface microbiome
  4. Adverse events
  5. Change in safety bloods, vital signs, FBC, renal function, CRP, LFTs
  6. Wound status (clinical infection, area, depth, extent of surface slough, pain by VAS, peri ulcer appearance)
  7. Patient well-being using a Visual Analogue Scale, 0-100mm.
  8. Vital signs (Resting pulse and blood pressure (BP))
Work Package 2: Safety of phage gel and overt toxic effect of phage gel. | 7 months
  The following outcomes will be recorded at weekly intervals for 4 weeks from baseline:
  1. change in surface microbiome
  2. Number of antibiotic-free days
  3. Adverse events
  4. Change in safety bloods, vital signs, FBC, renal function, CRP, LFTs
  5. Wound status (clinical infection, area, depth, extent of surface slough, pain by VAS, peri ulcer appearance)
  6. Patient well-being using a Visual Analogue Scale, 0-100mm.
  7. Eradication of clinical evidence of the infection in the index ulcer at weeks 1, 2 and 3, and time to eradication
  8. Healing of all ulcers and time to healing
  9. Resting pulse and blood pressure (BP)
Work Package 2: Clinical benefit and patient well-being associated with adding phage gel to systemically chosen antibiotics compared to placebo in the management of mild or moderate infection. | 16 months
  The following outcomes will be recorded at weekly intervals for 4 weeks from baseline:
  1. change in surface microbiome
  2. Number of antibiotic-free days
  3. Adverse events
  4. Change in safety bloods, vital signs, FBC, renal function, CRP, LFTs
  5. Wound status (clinical infection, area, depth, extent of surface slough, pain by VAS, peri ulcer appearance)
  6. Patient well-being using a Visual Analogue Scale, 0-100mm.
  7. Eradication of clinical evidence of the infection in the index ulcer at weeks 1, 2 and 3, and time to eradication
  8. Healing of all ulcers and time to healing
  9. Resting pulse and blood pressure (BP)
Work Package 2: Impact on the bacterial microbiome of systemically chosen antibiotics and of anti-staphylococcal phage gel. | 16 months
  The following outcomes will be recorded at weekly intervals for 4 weeks from baseline:
  1. change in surface microbiome
  2. Number of antibiotic-free days
  3. Adverse events
  4. Change in safety bloods, vital signs, FBC, renal function, CRP, LFTs
  5. Wound status (clinical infection, area, depth, extent of surface slough, pain by VAS, peri ulcer appearance)
  6. Patient well-being using a Visual Analogue Scale, 0-100mm.
  7. Eradication of clinical evidence of the infection in the index ulcer at weeks 1, 2 and 3, and time to eradication
  8. Healing of all ulcers and time to healing
  9. Resting pulse and blood pressure (BP)
Work Package 3: Safety of phage gel and overt toxic effect of phage gel. | 16 months
  The following outcomes will be recorded at weekly intervals for 4 weeks from baseline:
  1. Change in surface microbiome
  2. Number of antibiotic-free days
  3. Adverse events
  4. Change in safety bloods, FBC, renal function, CRP, LFTs
  5. Wound status (clinical infection, area, depth, extent of surface slough, pain by VAS, peri ulcer appearance)
  6. Patient well-being using a Visual Analogue Scale, 0-100mm.
  7. Eradication of clinical evidence of the infection in the index ulcer at weeks 1, 2 and 3, and time to eradication
  8. Healing of all ulcers and time to healing
  9. Resting pulse and blood pressure (BP)
Work Package 3: Clinical benefit and patient well-being associated with phage gel therapy compared to systemically chosen antibiotics in the management of mild infection. | 16 months
  The following outcomes will be recorded at weekly intervals for 4 weeks from baseline:
  1. Change in surface microbiome
  2. Number of antibiotic-free days
  3. Adverse events
  4. Change in safety bloods, FBC, renal function, CRP, LFTs
  5. Wound status (clinical infection, area, depth, extent of surface slough, pain by VAS, peri ulcer appearance)
  6. Patient well-being using a Visual Analogue Scale, 0-100mm.
  7. Eradication of clinical evidence of the infection in the index ulcer at weeks 1, 2 and 3, and time to eradication
  8. Healing of all ulcers and time to healing
  9. Resting pulse and blood pressure (BP)
Work Package 3: Impact on the bacterial microbiome of systemically chosen antibiotics and of anti-staphylococcal phage gel. | 16 months
  The following outcomes will be recorded at weekly intervals for 4 weeks from baseline:
  1. Change in surface microbiome
  2. Number of antibiotic-free days
  3. Adverse events
  4. Change in safety bloods, FBC, renal function, CRP, LFTs
  5. Wound status (clinical infection, area, depth, extent of surface slough, pain by VAS, peri ulcer appearance)
  6. Patient well-being using a Visual Analogue Scale, 0-100mm.
  7. Eradication of clinical evidence of the infection in the index ulcer at weeks 1, 2 and 3, and time to eradication
  8. Healing of all ulcers and time to healing
  9. Resting pulse and blood pressure (BP)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Derby and Burton NHS Foundation Trust, Derby, Derbyshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided